CLINICAL TRIAL: NCT02204410
Title: A Pilot Study of Omega-3 Fatty Acid Supplementation to ADHD Medication in Children With ADHD and Deficits in Emotional Self-Regulation
Brief Title: Omega-3 Supplementation to ADHD Medication in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Timothy Wilens, MD, Senior Staff, Pediatric Psychopharmaoclogy and Adult ADHD Clinic and Research Program; Associate professor of Psychiatry, Harvard Medical School; Director, Center for Addiction Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-P-000015
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-05

CONDITIONS: Attention Deficit Hyperactivity Disorder; Deficient Emotional Self-Regulation
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; DESR; Deficient Emotional Self-Regulation; Emotional Dysregulation; Omega-3 Fatty Acids; Fish Oil
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Fatty Acids, Omega-3; Fish Oils; Central Nervous System Stimulants; Methylphenidate; Dexmethylphenidate Hydrochloride; Lisdexamfetamine Dimesylate; Adderall; Dextroamphetamine; Amphetamine; Guanfacine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega-3 Fatty Acids and Stimulant Treatment (Experimental): Participants will receive open-label treatment with Omega-3 Fatty Acids. All participants must also be treated with a stable dose of a traditional ADHD medication at the time of enrollment.
  Interventions: Dietary Supplement: Omega-3 Fatty Acid; Drug: ADHD Medication

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acid
  Other Names: Fish Oil; Nordic Naturals Pro-Omega Junior Omega-3 Fatty Acid; Nordic Omega-3 Fishies
Drug: ADHD Medication
  Other Names: Stimulant; Concerta; Ritalin; Focalin; Vyvanse; Adderall; Dexedrine; Amphetamine; Methylphenidate; Stratterra; Tenex

SUMMARY:
This study is a 12-week open-label trial to assess the effectiveness of Omega-3 fatty acids for deficient emotional self-regulation (DESR) as a supplement to Attention Deficit/Hyperactivity Disorder (ADHD) treatment in children and adolescents with Attention Deficit/Hyperactivity Disorder. Subjects will be between the ages of 6-17 and will currently be on medication for their Attention Deficit/Hyperactivity Disorder but still experience DESR traits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children ages 6-17 years
* Living at home
* A diagnosis of ADHD (inattentive, hyperactive/impulsive, or combined type) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) based on clinical assessment
* Having a score outside the normal (a T-score of 60 or greater) on the Emotional Control subscale of the Behavior Rating Inventory of Executive Function (parent-report version) or a score outside the normal range (cumulative of 180 or greater) on the Anxious/Depressed, Attention Problems, and Aggressive Behavior subscales of the Child Behavior Checklist for ages (6-18)
* Currently on FDA approved traditional stimulant medication (such as Concerta of Adderall XR) or non-stimulant medication (such as Strattera or Tenex) for their ADHD for at least one month
* Beings able to come to weekly/monthly study visits for 12 weeks
* Having a parent or guardian with a level of understanding of the study

Exclusion Criteria:

* Having unstable medical illness as determined by the clinician investigator
* Having a current diagnosis of schizophrenia or bipolar disorder
* Having delusions or hallucinations
* Having a bleeding disorder
* Taking any other ongoing non-ADHD psychotropic medications other than stable, effective serotonin reuptake inhibitors such as fluoxetine (Prozac), citalopram (Celexa) or medications used on an as-needed basis
* Pregnant or nursing females
* IQ < 70 by previous testing or as judged by the clinician investigator
* Illegal substance use
* Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild
* Presence of suicidal risk, or homicidality
* Unwilling/unable to comply with study procedures
* Allergies to fish or shellfish or omega 3 fish oils; multiple adverse drug reactions
* Poor command of the English language

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E. Wilens, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: IRB-approved flyers were posted in the general community and throughout Massachusetts General Hospital between June 2014 and April 2016.
Period: Overall Study
Arm/Group | Omega-3 Fatty Acids and Stimulant Treatment
Started | 21
Completed | 10
Not Completed | 11
Not completed — Lost to Follow-up | 5
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Omega-3 Fatty Acids and Stimulant Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Emotional Control Subscale of the Behavior Rating Inventory of Executive Function - Parent Form (BRIEF-Parent)
Description: The Behavior Rating Inventory of Executive Function - Parent Form (BRIEF-Parent) is a 75-item checklist with a large normative sample, internal consistency, test-retest reliability, inter-rater reliability, and external and concurrent validity, divided into nine empirically and theoretically derived and T-scored subscales. The Emotional Control subscale measures the impact of executive function problems on emotional expression and assesses a child's ability to modulate or control his or her emotional responses. It is a 10-item subscale, and each item is scored "Never," "Sometimes," or "Often." Raw scores for all scales are computed with Software Portfolio (BRIEF-SP), which provides a raw score and T score (based on child's age) for each scale. Higher scores represent more greater emotional dysregulation.
Time Frame: Baseline and 12 Weeks
Population: Ten participants completed at least 6 weeks of the 12 week trial. These 10 participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3 Fatty Acids and Stimulant Treatment
Number analyzed (Participants) | 10
units on a scale
  Emotional Control Subscale T Score Baseline | 65.3 (10.2)
  Emotional Control Subscale T Score Endpoint | 58.4 (13.0)

2. Primary Outcome: Clinical Global Impression (CGI) Improvement for Deficient Emotional Self-Regulation (DESR)
Description: The Clinical Global Impression (CGI) is a clinician rated measure of illness severity, improvement, and efficacy of treatment (collected at all study visits). We examined the CGI Improvement specifically. The CGI Improvement for Deficient Emotional Self-Regulation (DESR) was reported at baseline and completion. The CGI-I is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. It is rated as:
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
Time Frame: Baseline and 12 Weeks
Population: Ten participants completed at least 6 weeks of the 12 week trial. These 10 participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3 Fatty Acids and Stimulant Treatment
Number analyzed (Participants) | 10
units on a scale
  CGI Improvement for DESR Baseline | 4.6 (0.7)
  CGI Improvement for DESR Endpoint | 3.0 (0.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from 10/1/2014 to 6/1/2016.
Description: Twelve subjects began taking taking open-label treatment with Omega-3 Fatty Acids. All of these subject's are included in adverse event reporting.
  Ten participants completed a minimum of 6 weeks of the 12 week trial. These 10 participants are included in the data analysis.
Arm/Group | Omega-3 Fatty Acids and Stimulant Treatment
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Fatty Acids and Stimulant Treatment (N=12)
Agitated/Tearful (Psychiatric disorders) | 2 (2)
Cold/Infection/Allergy (General disorders) | 3 (4)
Decreased Energy (Psychiatric disorders) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Increased Anxiety (Psychiatric disorders) | 1 (1)
Weight Gain/Increased Appetite (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No